CLINICAL TRIAL: NCT04655716
Title: Urine Alkalinisation to Prevent Acute Kidney Injury in COVID-19
Brief Title: Urine Alkalinisation to Prevent AKI in COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 283852
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate (Experimental): Intravenous sodium bicarbonate infusion
  Interventions: Drug: Sodium Bicarbonate 150Meq/L/D5W Inj
- Standard care (No Intervention): Standard of care by the clinical team

INTERVENTIONS:
Drug: Sodium Bicarbonate 150Meq/L/D5W Inj — Urine alkalinisation will be performed to achieve urine pH 7.5-8.5. Urine alkalinisation will be continued for up to 10 days or until patient is discharged or until primary endpoint is reached. Urine pH will be measured at point of care by dipstick.
  Other Names: 8.4% sodium bicarbonate intravenous form
  Arms: Sodium bicarbonate

SUMMARY:
The aim is to explore the feasibility and safety of urine alkalinisation in critically ill patients with COVID-19.

DETAILED DESCRIPTION:
Severe acute kidney injury appears to a major part of the SARS-CoV-2 syndrome. Preventing early acute kidney injury may reduce severe AKI as the disease progresses. Urine alkalinisation to prevent binding of SARS-COV-2 to renal tubular epithelial cells is a novel concept that could be used to design other therapies to reduce viral binding. Showing feasibility with this safe and available strategy could be the first step toward other related efforts.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Covid-19 positive
* Admission to Critical Care Unit
* Bladder catheter in situ
* Central line in place (including PICC line)
* Age ≥18y
* Written informed consent to participate in the study

Exclusion Criteria:

* Stage 3 AKI (as defined by KDIGO criteria)
* Chronic kidney disease stage 4 or 5
* Contraindications to NaHCO3 therapy (e.g. risk of serious drug interaction, systemic metabolic alkalosis, congestive heart failure)
* Urine pH > 7.0
* Serum sodium >150mmol/L
* Blood pressure >180/100mgHg
* Severe hypokalaemia (K<3.0mmol/L)
* Inability to grant informed consent
* Severe hypocalcaemia (Cai <0.8 mmol/L)
* Pregnant or lactating and breast-feeding women
* Unwilling to use contraception
* Patient is on a medication that may interact with sodium bicarbonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of patients treated who achieve >50% of urine measurements above pH 7.0 over the duration of intervention | up to 10 days after intensive care unit admission
  proportion of patients treated who achieve >50% of urine measurements above pH 7.0 over the duration of intervention

SECONDARY OUTCOMES:
number of days alive and free of stage 2-3 AKI (up to day 28) in each group | up to day 28 after randomisation
  number of days alive and free of stage 2-3 AKI (up to day 28) in each group
proportion of patients developing stage 2-3 AKI | up to day 28 after randomisation
  proportion of patients developing stage 2-3 AKI (or stage 3 if already at stage 2 at enrollment)
ventilator-free days | up to day 28 after randomisation
  ventilator-free days
hospital-free days | up to day 60 after randomisation
  hospital-free days

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No